

## EMPHASIS-lung ETOP 3-12

A randomized phase III trial of erlotinib versus docetaxel in patients with advanced squamous cell non-small cell lung cancer who failed first line platinum-based doublet chemotherapy stratified by VeriStrat Good vs VeriStrat Poor

Erlotinib Maldi TOF Phase III Signature in Squamous cell non-small cell lung cancer

A clinical trial of ETOP

## NCT01652469

| SAP VERSION | V.1 |
|-----------------------------|-----------------------------|
| SAP VERSION DATE | 07.01.2015 |
| TRIAL STATISTICIAN | Urania Dafni |
| TRIAL PRIMARY INVESTIGATORS | Egbert Smit, Solange Peters |
| DSMB SAP AUTHOR | Marie Kassapian |

 Table 1: Accrual by center

| Center | n (%) |
|-----------------------------------------------------------|------------|
| BEL063 Institut Jules Bordet, Brussels | xxx (xx.x) |
| CHE005 University Hospital Zürich, Zürich | xxx (xx.x) |
| CHE021 Centre Hospitalier Universitaire Vaudois, Lausanne | xxx (xx.x) |
| CHE022 Kantonsspital Luzern, Luzern | xxx (xx.x) |
| CHE024 Onkologiezentrum Thun - Berner Oberland, Thun | xxx (xx.x) |
| CHE105 Kantonsspital Graubünden, Chur | xxx (xx.x) |
| DNK003 Aarhus University Hospital, Aarhus | xxx (xx.x) |
| ESP052 Hospital Universitario 12 Octubre, Madrid | xxx (xx.x) |
| | xxx (xx.x) |
| | xxx (xx.x) |
| Total | XXX |

**Table 2:** Balance of treatment allocation per stratification factor combination

| | VeriStrat s | trat status=Good VeriStrat status= | | | tatus=Poor | | |
|---|---|---|---|---|---|---|---|
| PS=0&1 | | PS | =2 | 2 PS=0&1 | | | =2 |
| Treatment | Treatment | Treatment | Treatment | Treatment | Treatment | Treatment | Treatment |
| A | В | A | В | A | В | A | В |
| xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) | xxx (xx.x%) |

 Table 3a: Patient baseline characteristics (N=xx)

| Categorical characteristics | |
|---|---|
| Gender - n (%) | |
| Male | xxx (xx.x) |
| Female | xxx (xx.x) |
| Smoking history - n (%) | |
| Never | xxx (xx.x) |
| Former (>=100 cig & >=12 months smoke-free) | xxx (xx.x) |
| Current | xxx (xx.x) |
| Unknown | xxx (xx.x) |
| Histology - n (%) | |
| Squamous | xxx (xx.x) |
| Predominantly squamous with minor adenocarcinoma component | xxx (xx.x) |
| Predominantly squamous with adenocarcinoma component>10% | xxx (xx.x) |
| Unknown | xxx (xx.x) |
| Performance status - n (%) | |
| 0 | xxx (xx.x) |
| 1 | xxx (xx.x) |
| 2 | xxx (xx.x) |
| Veristrat status - n (%) | |
| Good | xxx (xx.x) |
| Poor | xxx (xx.x) |
| Continuous characteristics | |
| Age (yrs) | |
| Mean (95% CI) | xx.x (xx.x, xx.x) |
| Median (Min-Max) | xx.x (xx.x - xx.x) |

**Table 3b:** Patient baseline characteristics by treatment arm (N=xx)

| | Treatment A (n=37) | Treatment B (n=40) |
|---|---|---|
| Categorical charac | teristics | |
| Gender - n (%) | | |
| Male | xxx (xx.x) | xxx (xx.x) |
| Female | xxx (xx.x) | xxx (xx.x) |
| Smoking history - n (%) | | |
| Never | xxx (xx.x) | xxx (xx.x) |
| Former (≥100 cig & ≥12 months smoke-free) | xxx (xx.x) | xxx (xx.x) |
| Current | xxx (xx.x) | xxx (xx.x) |
| Unknown | xxx (xx.x) | xxx (xx.x) |
| Histology - n (%) | | |
| Squamous | xxx (xx.x) | xxx (xx.x) |
| Predominantly squamous with minor adenocarcinoma component | xxx (xx.x) | xxx (xx.x) |
| Predominantly squamous with adenocarcinoma component>10% | xxx (xx.x) | xxx (xx.x) |
| Unknown | xxx (xx.x) | xxx (xx.x) |
| Performance status - n (%) | | |
| 0 | xxx (xx.x) | xxx (xx.x) |
| 1 | xxx (xx.x) | xxx (xx.x) |
| 2 | xxx (xx.x) | xxx (xx.x) |
| Veristrat status - n (%) | | |
| Good | xxx (xx.x) | xxx (xx.x) |
| Poor | xxx (xx.x) | xxx (xx.x) |
| Continuous charac | teristics | |
| Age (yrs) | | |
| Mean (95% CI) | xx.x (xx.x, xx.x) | xx.x (xx.x, xx.x) |
| Median (Min-Max) | xx.x (xx.x - xx.x) | xx.x (xx.x - xx.x) |

Table 4a: Time on follow-up & time on treatment (N=xxx)

| Time on follow-up (in months) | All pts (xxx) |
|-------------------------------|--------------------|
| No. of pts still on f-up (%) | xxx (xx.x) |
| Median (Interq. Range) | xx.x (xx.x - xx.x) |
| Time-on treatment (in months) | |
| No. of discontinuations (%) | xxx (xx.x) |
| Median (Interq. Range) | xx.x (xx.x - xx.x) |

**Table 4b:** Time on follow-up & time on treatment by treatment arm (N=xxx)

| Time on follow-up (in months) | Treatment A<br>(n=xxx) | Treatment B<br>(n=xxx) |
|---|---|---|
| No. of pts still on f-up (%) | xxx (xx.x) | Xxx (xx.x) |
| Median (Interq. Range) | xx.x (xx.x - xx.x) | xx.x (xx.x - xx.x) |
| Time-on treatment (in months) | | |
| No. of discontinuations (%) | xxx (xx.x) | xxx (xx.x) |
| Median (Interq. Range) | xx.x(xx.x - xx.x) | xx.x (xx.x - xx.x) |

**Table 5a:** Adverse event overview

| | N | % |
|----------------|-----|------|
| Experienced AE | XXX | XX.X |
| No AE | XXX | XX.X |
| Total subjects | XXX | |

**Table 5b:** Adverse event overview by treatment arm

| | Treati | Treatment A | | nent B |
|----------------|--------|-------------|-----|--------|
| | N | % | N | % |
| Experienced AE | XXX | XX.X | XXX | XX.X |
| No AE | XXX | XX.X | XXX | XX.X |
| Total subjects | XXX | | XXX | |

 Table 6a: Serious adverse event overview

| | N | % |
|-----------------|-----|------|
| Experienced SAE | XXX | XX.X |
| No SAE | XXX | XX.X |
| Total subjects | XXX | |

Table 6b: Serious adverse event overview by treatment arm

| | Treati | ment A | Treatment B | |
|-----------------|---------|--------|-------------|------|
| | N | % | N | % |
| Experienced SAE | XXX | XX.X | XXX | XX.X |
| No SAE | XXX | XX.X | XXX | XX.X |
| Total subjects | XXX XXX | | XXX | |

**Table 7:** Serious adverse events overview by center

| Center | No. of patients | Experienced<br>SAE | | <u>-</u> | | Total<br>follow-up | SAE<br>incidence |
|---|---|---|---|---|---|---|---|
| | 1 | N | % | (months) | | | |
| BEL063 Institut Jules Bordet | XXX | XXX | XX.X | XX.X | XX.X | | |
| CHE005 University Hospital Zürich | XXX | XXX | XX.X | XX.X | XX.X | | |
| CHE021 Centre Hospitalier Universitaire Vaudois | XXX | XXX | XX.X | XX.X | XX.X | | |
| CHE022 Kantonsspital Luzern | XXX | XXX | XX.X | XX.X | XX.X | | |
| CHE024 Onkologiezentrum Thun - Berner<br>Oberland | XXX | XXX | XX.X | XX.X | xx.x | | |
| CHE105 Kantonsspital Graubünden | XXX | XXX | XX.X | XX.X | XX.X | | |
| DNK003 Aarhus University Hospital | xxx | XXX | XX.X | XX.X | XX.X | | |
| ESP052 Hospital Universitario 12 Octubre | xxx | XXX | XX.X | XX.X | XX.X | | |
| ESP055 Hospital General Universitario Alicante | xxx | XXX | XX.X | XX.X | XX.X | | |
| | xxx | XXX | XX.X | XX.X | XX.X | | |
| | XXX | XXX | XX.X | XX.X | XX.X | | |

 Table 8a: Frequency of serious adverse events

| Adverse event description | Total |
|------------------------------------------------|-------|
| Febrile neutropenia | XXX |
| Pain | XXX |
| Respiratory failure | XXX |
| Respiratory, thoracic and mediastinal disorder | XXX |
| Bronchial infection | XXX |
| Bronchial obstruction | XXX |
| Bronchopulmonary hemorrhage | XXX |
| | XXX |
| | XXX |
| Total | XXX |

**Table 8b:** Frequency of serious adverse events by treatment arm

| Adverse event description | Treatment A | Treatment B | Total |
|-----------------------------|-------------|-------------|-------|
| Bronchial infection | xxx (xx.x) | xxx (xx.x) | XXX |
| Bronchial obstruction | xxx (xx.x) | xxx (xx.x) | XXX |
| Bronchopulmonary hemorrhage | xxx (xx.x) | xxx (xx.x) | XXX |
| Dehydration | xxx (xx.x) | xxx (xx.x) | XXX |
| Endocrine disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| Febrile neutropenia | xxx (xx.x) | xxx (xx.x) | XXX |
| Fever | xxx (xx.x) | xxx (xx.x) | XXX |
| Gastrointestinal disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | XXX |
| Total | XXX | XXX | XXX |

**Table 9a:** Frequency of serious adverse events according to CTCAE Version 4

| Adverse event description | Total | % |
|------------------------------------------------------|-------|------|
| Respiratory, thoracic and mediastinal disorders | XXX | XX.X |
| General disorders and administration site conditions | XXX | XX.X |
| Blood and lymphatic system disorders | XXX | XX.X |
| Infections and infestations | XXX | XX.X |
| Endocrine disorders | XXX | XX.X |
| Gastrointestinal disorders | XXX | XX.X |
| | XXX | XX.X |
| | XXX | XX.X |
| Total | XXX | |

**Table 9b:** Frequency of serious adverse events by treatment arm according to CTCAE Version 4

| Adverse event description | Treatment A | Treatment B | Total |
|---|---|---|---|
| Blood and lymphatic system disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| Endocrine disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| Gastrointestinal disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| General disorders and administration site conditions | xxx (xx.x) | xxx (xx.x) | XXX |
| Infections and infestations | xxx (xx.x) | xxx (xx.x) | XXX |
| Injury, poisoning and procedural complications | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | XXX |
| Total | XXX | XXX | xxx |

**Table 10:** Number of patients experiencing specific number of serious adverse events

| | SAEs | | |
|-------------------|------|-----|-----|
| Frequency of SAEs | 1 | 2 | 3 |
| No. of patients | XXX | XXX | XXX |

**Table 11:** Number of patients experiencing specific number of serious adverse events according to CTCAE Version 4

| | SAEs | | |
|-------------------|------|-----|-----|
| Frequency of SAEs | 1 | 2 | 3 |
| No. of patients | xxx | XXX | XXX |

**Table 12:** Distribution of adverse events by Grade

| Adverse event description | Grade=1 | Grade=2 | Grade=3 | Grade=4 | Grade=5 | Total |
|---|---|---|---|---|---|---|
| Abdominal distension | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Abdominal pain | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Alanine aminotransferase increase | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Allergic rhinitis | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Alopecia | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Amnesia | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Anemia | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Total | XXX | xxx | xxx | xxx | xxx | XXX |

**Table 13:** Distribution of adverse events by Grade according to CTCAE Version 4

| Adverse event description | Grade=1 | Grade=2 | Grade=3 | Grade=4 | Grade=5 | Total |
|---|---|---|---|---|---|---|
| Blood and lymphatic system disorders | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Cardiac disorders | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Endocrine disorders | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Eye disorders | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Gastrointestinal disorders | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Hepatobiliary disorders | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Infections and infestations | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | xxx (xx.x) | XXX |
| Total | XXX | xxx | xxx | xxx | XXX | XXX |

 Table 14a: Frequency of adverse events

| Adverse event description | Total | Adverse event description | Total |
|----------------------------|-------|---------------------------|-------|
| Fatigue | XXX | Amnesia | XXX |
| Rash maculo papular | XXX | Anemia | XXX |
| Dyspnea | XXX | Back pain | XXX |
| Cough | xxx | Bronchial obstruction | XXX |
| Diarrhea | XXX | Bronchospasm | XXX |
| Mucositis oral | XXX | Death NOS | XXX |
| Anorexia | XXX | Dehydration | XXX |
| Febrile neutropenia | xxx | Dry mouth | XXX |
| Neutrophil count decreased | XXX | Endocrine disorders | XXX |
| | XXX | | XXX |

**Table 14b:** Frequency of adverse events by treatment arm

| Adverse event description | Treatment A | Treatment B | Total |
|-----------------------------------|-------------|-------------|-------|
| Abdominal distension | xxx (xx.x) | xxx (xx.x) | XXX |
| Abdominal pain | xxx (xx.x) | xxx (xx.x) | XXX |
| Alanine aminotransferase increase | xxx (xx.x) | xxx (xx.x) | XXX |
| Allergic rhinitis | xxx (xx.x) | xxx (xx.x) | XXX |
| Alopecia | xxx (xx.x) | xxx (xx.x) | XXX |
| Amnesia | xxx (xx.x) | xxx (xx.x) | XXX |
| Anemia | xxx (xx.x) | xxx (xx.x) | XXX |
| Anorexia | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | XXX |
| Total | xxx | XXX | xxx |

**Table 15a:** Frequency of adverse events according to CTCAE Version 4

| Adverse event description | Total | % |
|------------------------------------------------------|-------|------|
| General disorders and administration site conditions | xxx | XX.X |
| Skin and subcutaneous tissue disorders | xxx | XX.X |
| Respiratory, thoracic and mediastinal disorders | xxx | XX.X |
| Gastrointestinal disorders | xxx | XX.X |
| Blood and lymphatic system disorders | xxx | XX.X |
| Infections and infestations | xxx | XX.X |
| | xxx | XX.X |
| | XXX | XX.X |
| Total | XXX | |

| Adverse event description | Treatment A | Treatment B | Total |
|---|---|---|---|
| Blood and lymphatic system disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| Cardiac disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| Endocrine disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| Eye disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| Gastrointestinal disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| General disorders and administration site conditions | xxx (xx.x) | xxx (xx.x) | XXX |
| Hepatobiliary disorders | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | XXX |
| | xxx (xx.x) | xxx (xx.x) | XXX |
| Total | xxx | xxx | XXX |

**Table 16:** Number of patients experiencing specific number of adverse events

| | AEs | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Frequency of AEs | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 |
| No. of patients | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | xxx | XXX | XXX | XXX |

**Table 17:** Number of patients experiencing specific number of adverse events according to CTCAE Version 4

| | | | | | | | AEs | | |
|------------------|-----|-----|-----|-----|-----|-----|-----|-----|-----|
| Frequency of AEs | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 |
| No. of patients | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX | XXX |

 Table 18a: Frequency of targeted adverse events

| Adverse event description | N | % |
|-----------------------------------|-----|------|
| Fatigue | XXX | XX.X |
| Rash maculo papular | XXX | XX.X |
| Dyspnea | XXX | XX.X |
| Diarrhea | XXX | XX.X |
| Mucositis oral | XXX | XX.X |
| Neutrophil count decreased | XXX | XX.X |
| Febrile neutropenia | XXX | XX.X |
| Alanine aminotransferase increase | XXX | XX.X |
| Pain | XXX | XX.X |
| Peripheral sensory neuropathy | XXX | XX.X |
| | XXX | XX.X |
| | XXX | XX.X |
| Total | xxx | |

**Table 18b:** Frequency of non-targeted adverse events

| Adverse event description | N | % | Adverse event description | N | % |
|---|---|---|---|---|---|
| Cough | xxx | XX.X | Fatigue | XXX | XX.X |
| Anorexia | xxx | XX.X | Gastrointestinal disorders | XXX | XX.X |
| Alopecia | xxx | XX.X | Glucose intolerance | XXX | XX.X |
| Pain | xxx | XX.X | Hepatic pain | XXX | XX.X |
| Conjunctivitis | xxx | XX.X | Hypertriglyceridemia | XXX | XX.X |
| Constipation | XXX | XX.X | Hyponatremia | XXX | XX.X |
| Dizziness | xxx | XX.X | Infections and infestations | XXX | XX.X |
| Lung infection | xxx | XX.X | Keratitis | XXX | XX.X |
| Nausea | XXX | XX.X | Laryngeal hemorrhage | XXX | XX.X |
| Abdominal pain | XXX | XX.X | Leukocytosis | XXX | XX.X |
| Bone pain | xxx | XX.X | Mucosal infection | XXX | XX.X |
| Creatinine increased | xxx | XX.X | Mucositis oral | XXX | XX.X |
| Total=vvv | | | | | |

Total=xxx

**Table 19a:** Frequency of targeted adverse events according to CTCAE Version 4

| Adverse event description | N | % |
|------------------------------------------------------|-----|------|
| General disorders and administration site conditions | xxx | XX.X |
| Skin and subcutaneous tissue disorders | XXX | XX.X |
| Respiratory, thoracic and mediastinal disorders | XXX | XX.X |
| Blood and lymphatic system disorders | XXX | XX.X |
| Gastrointestinal disorders | XXX | XX.X |
| Infections and infestations | XXX | XX.X |
| Investigations | XXX | XX.X |
| | XXX | XX.X |
| | XXX | XX.X |
| Total | xxx | |

**Table 19b:** Frequency of non-targeted adverse events according to CTCAE Version 4

| Adverse event description | N | % |
|------------------------------------------------------|-----|------|
| Gastrointestinal disorders | XXX | XX.X |
| Respiratory, thoracic and mediastinal disorders | XXX | XX.X |
| Skin and subcutaneous tissue disorders | XXX | XX.X |
| Metabolism and nutrition disorders | XXX | XX.X |
| General disorders and administration site conditions | XXX | XX.X |
| Musculoskeletal and connective tissue disorders | XXX | XX.X |
| Nervous system disorders | XXX | XX.X |
| Eye disorders | XXX | XX.X |
| | XXX | XX.X |
| | XXX | XX.X |
| Total | xxx | |

Table 20a: Treatment A: Adverse event information by patient (any AE & SAE)

| ID | Adverse event<br>(CTCAE V.4) | Adverse event description | AE/<br>SAE | Grade | Date of onset | Relate<br>d cycle | Relation to treatment | Outcome |
|---|---|---|---|---|---|---|---|---|
| 4101 | Respiratory, thoracic and mediastinal disorders | Allergic rhinitis | AE | 2 | | 2 | 4-probable | |
| | Metabolism and nutrition disorders | Anorexia | AE | 2 | | 4 | 3-possible | PD (15/04/2013) |
| | Respiratory, thoracic and mediastinal disorders | Bronchospasm | AE | 1 | | 4 | 1-unrelated | & Death |
| | Eye disorders | Conjunctivitis | AE | 1 | | 4 | 3-possible | (26/09/2013) |
| | Skin and subcutaneous tissue disorders | Rash maculo<br>papular | AE | 2 | 01/02/2013 | 4 | 5-definite | |
| 4243 | Skin and subcutaneous tissue disorders | Rash maculo<br>papular | AE | 2 | 17/04/2013 | 1 | 5-definite | |
| | Respiratory, thoracic and mediastinal disorders | Cough | AE | 2 | | 3 | 1-unrelated | On Fallow up |
| | Metabolism and nutrition disorders | Anorexia | AE | 3 | | 4 | 3-possible | On Follow-up |
| | Musculoskeletal and connective tissue disorders | Back pain | AE | 1 | | 4 | 1-unrelated | |

**Table 20b:** Treatment B: Adverse event information by patient (any AE & SAE)

| ID | Adverse event (CTCAE V.4) | Adverse event description | AE/<br>SAE | Grad<br>e | Date of onset | Relate<br>d cycle | Relation to treatment | Outcome |
|---|---|---|---|---|---|---|---|---|
| 4270 | General disorders and administration site conditions | Fatigue | AE | 1 | 09/05/2013 | 2 | 3-possible | PD (19/09/2013) |
| | Skin and subcutaneous tissue disorders | Alopecia | AE | 2 | | 3 | 5-definite | &<br>Death |
| | Nervous system disorders | Amnesia | AE | 2 | | 3 | 1-unrelated | (30/11/2013) |
| | Vascular disorders | Hypertension | AE | 2 | | 3 | 3-possible | |
| 4411 | Blood and lymphatic<br>system disorders | Febrile<br>neutropenia | SAE | 4 | 10/05/2013 | 1 | 5-definite | Death (30/05/2013) |
| 4413 | Infections and infestations | Bronchial<br>infection | SAE | 3 | 15/06/2013 | 2 | 3-possible | On Fallow up |
| | Infections and infestations | Sensis | | 4 | 27/06/2013 | 2 | 5-definite | On Follow-up |

 Table 21: Narratives of patients with a SAE

| ID | SAE | Date of onset | Narrative |
|---|---|---|---|
| 4411 | Febrile neutropenia | 10/05/2013 | 63 year old formerly smoking man with medical history of asthma and urothelial carcinoma (2009) was diagnosed with advanced, progressing (adrenal, bone, brain, liver and lung metastases) squamous cell NSCLC after surgery |
| 4413 | Bronchial infection | 15/06/2013 | 56 year old smoking man with medical history of hypertension and diabetes was diagnosed with advanced, progressing (liver and lymph node metastases) squamous cell NSCLC after radiotherapy and chemoradiotherapy |

**Table 22:** Adverse events experienced by patients with Progression of disease and/or Death

| | ID number | | | | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse event | 4101 | 4270 | 4290 | 4411 | 4432 | 4434 | 4435 | 4441 | 4442 | 4459 | 4461 | 4471 | 4475 | 4477 | 4496 | 4506 | 4509 | 4511 | 4515 |
| Allergic rhinitis | ✓ | | | | | | | | | | | | | | | | | | |
| Alopecia | | ✓ | | | | | | | | | | | | | | | | | |
| Amnesia | | ✓ | | | | | | | | | | | | | | | | | |
| Anorexia | ✓ | | | | 1 | | | | | ✓ | | | | | | | | | |
| Bone pain | | | | | | | | | | | | | ✓ | | | | | | |
| Bronchial infection | | | | | | | | | ✓ | | | | | | | | | | |

**Table 23:** Adverse events experienced by patients with Progression of disease and/or Death according to CTCAE Version 4

| | | | | | | | | | ID | numb | er | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse event | 4101 | 4270 | 4290 | 4411 | 4432 | 4434 | 4435 | 4441 | 4442 | 4459 | 4461 | 4471 | 4475 | 4477 | 4496 | 4506 | 4509 | 4511 | 4515 |
| Endocrine<br>disorders | | | | | | _ | | | | <del>-</del> | | | - | | ✓ | | | - | <del></del> |
| Eye disorders | ✓ | | | | | | | | | | | | | | | | | | |
| Gastrointestinal disorders | | | | | ✓ | | ✓ | ✓ | | | | | | | | ✓ | | ✓ | |
| Hepatobiliary<br>disorders | | | | | | | | | | | | | ✓ | | | | | | |
| Infections and infestations | | | ✓ | | | | | ✓ | 1 | | | | | | | | | | |
| Investigations | | | | | | | | | | | | | | | ✓ | | | ✓ | |